CLINICAL TRIAL: NCT02067091
Title: Performance of Bioresorbable Scaffold in Primary Percutaneous Intervention of ST Elevation Myocardial Infarct (BVS in STEMI)
Brief Title: Performance of Bioresorbable Scaffold in Primary Percutaneous Intervention of ST Elevation Myocardial Infarct
Acronym: BVS in STEMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Feiring (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/2006
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
Keywords: STEMI; Coronary; Bioresorbable scaffold; Drug eluting stent; Optical coherence tomography; Multislice computed tomography
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BVS (Active Comparator): Implantation of bioresorbable vascular scaffold in coronary artery by direct stenting after thrombus aspiration by percutaneous coronary intervention
  Interventions: Device: stent implant in a coronary artery
- DES (Active Comparator): Implantation of drug eluting stent in coronary artery by direct stenting after thrombus aspiration by percutaneous coronary intervention
  Interventions: Device: stent implant in a coronary artery

INTERVENTIONS:
Device: stent implant in a coronary artery — Implantation of device called a stent in a coronary artery
  Percutaneous coronary intervention

SUMMARY:
Patients presenting with acute ST elevation myocardial infarct urgently need revascularization. Standard of care is establishing bloodflow through the coronary vessels using thrombus aspiration catheter, and securing the result by using a metallic drug eluting stent. New kinds of non-metallic bioresorbable stents are now available. They have however challenges in structural strength.

The investigators want to compare the new bioresorbable scaffold with traditional metallic stents in this setting in a prospective, randomized, non-blinded, multicenter study in 120 patients. The investigators will use an imaging technique, optical coherence tomography, to evaluate the results after 12 months.

The investigators also want to see if modern multislice computed tomography can give useful information in the follow-up of stented coronary arteries after 12 and 24 months.

DETAILED DESCRIPTION:
Patients presenting with ST elevation myocardial infarction for primary PCI (percutaneous coronary intervention) will be screened. After thrombus aspiration, patient will be asked for oral consent if TIMI flow 2-3. Patient will then be randomized between drug eluting stent (Xience pro, Abbott Vascular Solutions) and bioresorbable scaffold (Absorb, Abbott Vascular Solutions). Optical coherence tomography (OCT) will be performed before stenting and after final result. Stent will be deployed without further predilatation if possible. Follow up at 12 months (clinical, angio with OCT and multislice CT coronary angiogram (MSCT-CA)) and 24 months (MSCT-CA).

ELIGIBILITY:
Inclusion Criteria:

1. History of chest pain < 12 hrs
2. ST elevation of ≥ 2 mm in ≥2 contiguous precordial leads (V1-V6), and/or ≥ 1 mm in ≥ 2 contiguous standard leads (I, II, III, aVf, aVr,aVl).
3. Clinical decision to treat with primary PCI
4. > 18 years
5. Oral informed consent

Exclusion Criteria:

1. Contraindications to long term double antiplatelet therapy
2. Known kidney failure with GFR < 45
3. Cardiac arrest or severe cardiogenic shock (Persistent BP <90 mmHg, despite adequate treatment)
4. Other severe illness with life expectancy of less than 12 months (eg. malignancy, severe malnutrition, degenerative disease)

Procedural contraindications:

1. Heavy calcification, tortuous vessel or large side branch (> 2,5 mm) at culprit lesion.
2. TIMI 0-1 flow after aspiration
3. Unable to advance thrombus aspiration catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Coronary Stent Healing Index (cumulated) | 12 months
  1. Uncovered struts: 2% =1 - 5% =2 - 10% =3 - 15% =4 - 20% =5 - 25% =6 - 30% =7 - 35% =8 - 40% =9
  2. Uncovered struts in front of side branch on acquired or persistent malposed struts. 10% =1 - 20% =2 - 30% =3 etc… til 100%=10
  3. Persistent malposition: ≥2 nabo struts længde mindst 1 mm =1 ; ≥2mm=3 ; ≥3 mm = 3
  4. Acquired malposition: ≥2 adjacent struts of at least 1 mm length =2 ; ≥2mm=4 ; ≥3 mm = 6
  5. Neointimal thickness in one frame >200 =1 - >300 =2 - >400 =3 or diameter stenosis >50% =4 - > 75% =5
  6. Cumulated extra stent lumen increase in match cross sectional analysis: (gns. areal mål): ≥0.2mm2 =1 ; ≥0.4 mm2 = 2; ≥0.6mm2=3 ; ≥0.8 mm2 = 4 ; ≥1.0 mm2=5 ; ≥1.2 mm2 = 6
Multislice computed tomography | 24 months
  MSCT-CA will be done at 24 months to extend the observational time by a non-invasive measure. MSCT-CA will be compared to conventional angiogram with OCT at 12 months to verify MSCT-CA findings at 24 months. Results will be reported in separate paper.
Minimum Flow Area | 12 months
  Minimum flow area as defined in TROFI I, measured by OCT

SECONDARY OUTCOMES:
Total Death | 5 years
  Total death encompasses cardiac death and other fatal categories, which include cerebrovascular death, death from other cardiovascular disease (i.e. pulmonary embolism, dissection aortic aneurysm will be included in this category), death from malignant disease, death from suicide, violence or accident, or death from other reasons.
Cardiac death | 5 years
  Cardiac death encompasses coronary heart disease death including fatal myocardial infarction, sudden cardiac death including fatal arrhythmias and cardiac arrest without successful resuscitation, death from heart failure including cardiogenic shock, and death related to a cardiac procedure or surgery within 28 days from the procedure.
Myocardial infarction | 5 years
  Evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Under these conditions any one of the following criteria meets the diagnosis for myocardial infarction :
  1. Detection of rise and/or fall of preferably troponin T with at least one value above the 99th percentile of the upper reference limit (URL) together with evidence of myocardial ischemia with at least one of the following (MI types 1 or 2):
     1. Symptoms of ischemia
     2. ECG changes indicative of new ischemia (new ST-T changes or new LBBB)
     3. Development of pathological Q waves in the ECG
     4. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality
  2. Sudden, unexpected cardiac death, involving cardiac arrest.
Stent thrombosis | 5 years
  Stent thrombosis is recognized when documented by angiography and/or autopsy and when meeting the criteria for spontaneous myocardial infarction occurring in the territory of the treated vessel (11). Stent thrombosis are categorized as acute, sub-acute, late and very late and as definite, probable and possible according to the ARC-criteria (12).
Target Lesion and vessel Revascularization | 5 years
  Coronary artery bypass grafting with grafting or PCI of index lesion. Coronary artery bypass grafting with grafting or PCI of index vessel.
Non Target vessel revascularisation | 5 years
  All PCI or coronary bypass grafting of non index vessel
Stable angina | 5 years
  Angina as reported by patient, classified according to Canadian cardiac society class (CCS)
Vascular cerebral events | 5 years
  Vascular events documented by neurological permanent disabilities or by diagnostic imaging (MRI or CT).
Admission for congestive heart failure or arrhythmias | 5 years
  Admissions were the diagnosis at release is one of heart failure or arrhythmias
Optical Coherence tomography | 12 months
  Area stenosis
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  TIMI flow pre and post PCI
Biochemical | 12 months
  Creatinine, hemoglobin, Troponin T will be analyzed during index procedure post procedure and at 12 months follow-up. ProBNP will be analyzed at 12 months follow-up
Markers | 12 months
  Plasma, full blood, serum and urine will be drawn immediately after the procedure and frozen in a bio bank for later analysis
Thrombus analysis | At index procedure were the patient is included and randomized
  Visible thrombus aspirates will be sent for analysis
Optical coherence tomography | 12 months
  Lumen late loss
Optical coherence tomography | 12 months
  Crushed stent segments
Optical coherence tomography | 12 months
  Malposition of stent segments
Optical coherence tomography | 12 months
  Minimum expansion of stent struts expressed as absolute area and percentage of closest reference reference area
Optical coherence tomography | 12 months
  Vessel ostial stented area (acute and at FU)
Optical coherence tomography | 12 months
  Thrombus burden
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Blush grade
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Thrombus burden
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Angiographic complications
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Contrast use
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Procedure time
Angiographic endpoints at index admission | After index procedure were the patient is included and randomized
  Radiation skin dose

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Tuseth, PhD, Study Chair — University of Bergen; Jan Erik Nordrehaug, PhD, Study Chair — University of Bergen; Erlend Eriksen, MD, Principal Investigator — Helse-Bergen HF
Locations (2):
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided